CLINICAL TRIAL: NCT03224234
Title: A Randomized Study to Evaluate the Efficacy of Insulclock® in Patients With Uncontrolled Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Insulcloud S.L. (Industry)
Responsible Party: Principal Investigator, Guillermo Umpierrez, MD, Professor of Medicine, Emory University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB00094393
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Diabetes
Keywords: Uncontrolled Type 2 Diabetes; Insulclock; Electronic device; Alarm system
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: At midpoint (week 12), patients will be converted to the alternate arm (cross-over design).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Insulclock with feedback (Group A) (Experimental): Participants will use the Insulclock and receive daily information on their smartphone on insulin administration (time and dosing) as well as reminders in the event of missing doses. At midpoint (week 12), patients will be converted to the alternate arm.
  Interventions: Device: Insulclock with feedback
- Insulclock without feedback (Group B) (Active Comparator): Participants will use the Insulclock, but will not receive feedback on insulin administration. At midpoint (week 12), patients will be converted to the alternate arm.
  Interventions: Device: Insulclock without feedback

INTERVENTIONS:
Device: Insulclock with feedback — Daily information on a smartphone on insulin administration (time and dosing) as well as reminders in the event of missing doses.
  Arms: Insulclock with feedback (Group A)
Device: Insulclock without feedback — Not feedback on insulin administration.
  Arms: Insulclock without feedback (Group B)

SUMMARY:
Poor adherence to insulin regimens is reported in up to two-third of patients with diabetes; thus it is important to identify patients at risk and to develop strategies and tools to increase adherence to prescribed insulin regimens. This study will evaluate the efficacy of Insulclock® - small electronic device to help track date, time and dosage of the last injection, type of insulin used and temperature, with an alarm system to prevent insulin omissions and mistiming.

DETAILED DESCRIPTION:
Diabetes is arguably the most urgent healthcare challenge of the 21st century. Poor adherence to insulin regimens is reported in up to two-third of patients with diabetes; thus it is important to identify patients at risk and to develop strategies and tools to increase adherence to prescribed insulin regimens. This study will evaluate the efficacy of Insulclock® - small electronic device to help track date, time and dosage of the last injection, type of insulin used and temperature, with an alarm system to prevent insulin omissions and mistiming. The Insulclock's real time memory and alert system are likely to improve treatment adherence, patient's satisfaction, and quality of life measures, which may improve glycemic control in insulin treated patients with Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 80 years
* Diagnosis of T2D
* Screening HbA1c ≥ 7.5% to ≤ 11%
* Continuous treatment with one or more oral antidiabetic agents, for at least 2 months
* Continuous treatment with daily basal insulin (NPH, glargine U100 or detemir), for at least 2 months, (insulin dose ≤0.5U/Kg/day)
* If patients are on combination therapy of basal insulin and GLP1-RA, the dose of GLP-1 RA should be stable for the past three months.
* Owns a smartphone - Apple iPhone, Samsung Galaxy models
* Signed, informed consent and HIPAA documentation
* Subjects' ability to self-administer insulin, use the device and complete subject reported outcomes instruments
* Subjects' ability & willingness to adhere to and be compliant with study protocol

Exclusion Criteria:

* Refusal or inability to give informed consent to participate in the study
* Subject is currently taking or was treated with glargine U300 insulin, degludec, insulin dose greater than 0.5 U/kg/day during the previous three months
* Subject treated with prandial insulin or premixed formulations during the previous three months
* Impaired renal function as shown by, but not limited to, eGFR < 30 ml/min.
* Muscle weakness or hemiparesis related to previous stroke or myelopathy resulting in incoordination, muscle weakness and inability to use pen device for insulin administration
* History of diabetic ketoacidosis during the previous 6 months
* Clinical evidence of active liver disease, or serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) 3 times the upper limit of the normal range
* History of hypoglycemia unawareness
* Pregnancy or lactation
* Known hypersensitivity to insulin glargine or any of the components
* Any malignancy within the last 5 years, except for adequately treated basal or squamous cell carcinoma of the skin or adequately treated cervical carcinoma in situ
* Current drug addiction or current alcohol abuse, or history of substance or alcohol abuse within the last 2 years
* Diagnosis of dementia
* Severe gastrointestinal diseases including gastroparesis
* Cardiac status NYHA III-IV
* Acute infection
* Patients on or planning to receive long term oral or injectable steroid treatment for greater than 10 days
* Patient schedule to undergo general surgery during the next 6 months
* Any disease or condition that in the opinion of the investigator and/or sponsor may interfere with the completion of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (1):
- Emory Clinic, Emory University Hospital (non-CRN), Emory University Hospital Clinical Research Network, Emory University Hospital Midtown, Grady Health System (non-CRN), Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consented 121 participants. The study team realized that changes needed to be done for the protocol to be efficient. The first 28 candidates were consented for "pilot" data, ten of them were screen failures, 18 were randomized. Data on Insulclock device malfunctions were collected, it was planned to improve all issues by the time the main phase of the study started. 93 subjects were consented for the main study, 13 were screen failures, and 80 subjects were randomized.
Period: Main Study
Arm/Group | Insulclock With Feedback (Group A) | Insulclock Without Feedback (Group B)
Started | 40 | 40
Completed | 35 | 35
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 5 | 5
Period: Pilot
Arm/Group | Insulclock With Feedback (Group A) | Insulclock Without Feedback (Group B)
Started | 11 | 7
Completed | 11 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pilot: Insulclock With Feedback (Group A): Participants use the Insulclock and receive daily information on their smartphone on insulin administration (time and dosing) as well as reminders in the event of missing doses. During the study period, information is collected on problems with connectivity, malfunction or any problem with the Insulclock® device.
- Pilot:Insulclock Without Feedback (Group B): Participants use the Insulclock, but will not receive feedback on insulin administration.
  During the study period, information is collected on problems with connectivity, malfunction or any problem with the Insulclock® device.
- Total: Total of all reporting groups
Arm/Group | Insulclock With Feedback (Group A) | Insulclock Without Feedback (Group B) | Pilot: Insulclock With Feedback (Group A) | Pilot:Insulclock Without Feedback (Group B) | Total
Number analyzed (Participants) | 40 | 40 | 11 | 7 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 35 | 35 | 11 | 7 | 88
  >=65 years | 5 | 5 | 0 | 0 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Main study phase: Female | 27 | 17 | 6 | 3 | 53
  Main study phase: Male | 13 | 23 | 5 | 4 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 36 | 37 | 11 | 6 | 90
  White | 1 | 3 | 0 | 0 | 4
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 0 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 11 | 7 | 98

OUTCOME MEASURES:

1. Primary Outcome: Number of Insulin Injection Irregularities.
Description: Number of insulin injection irregularities (omission, mistiming and dosing) will be registered on the Insulclock device, and data will be retrieved during each clinic visit to monitor treatment adherence.
Time Frame: Week 0 through week 24.
Population: Data were collected as a part of main phase of the study only.
Measure: Mean (Standard Deviation); unit: irregularities
Groups:
- Pilot: Insulclock Without Feedback (Group B): Participants use the Insulclock, but will not receive feedback on insulin administration.
  During the study period, information is collected on problems with connectivity, malfunction or any problem with the Insulclock® device.
Arm/Group | Insulclock With Feedback (Group A) | Insulclock Without Feedback (Group B) | Pilot: Insulclock With Feedback (Group A) | Pilot: Insulclock Without Feedback (Group B)
Number analyzed (Participants) | 40 | 40 | 0 | 0
irregularities | 22.22 (25.12) | 23.10 (26.75) |  |

2. Primary Outcome: Number of Participants Experiencing Insulclock Device Malfunctions
Description: Number of participants experiencing Insulclock device malfunctions are reported
Time Frame: Up to 12 weeks
Population: Data were collected as a part the pilot phase. Data on Insulclock device malfunctions were collected, it was planned to improve all issues by the time the main phase of the study started.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulclock With Feedback (Group A) | Insulclock Without Feedback (Group B) | Pilot: Insulclock With Feedback (Group A) | Pilot:Insulclock Without Feedback (Group B)
Number analyzed (Participants) | 0 | 0 | 11 | 7
Participants |  |  | 5 | 2

3. Secondary Outcome: Change in Diabetes Treatment Satisfaction Questionnaire (DTSQc-change) Score.
Description: The amplitude of the score on the DTSQc gives the degree of change in satisfaction while the direction (positive or negative) will provide guidance on the preference of one device over the other. DTSQc contains eight items scored on 7-point scales; scores range from +3 = much more satisfied now to -3 = much less satisfied now, with 0 (midpoint), representing no change.
Time Frame: Baseline, 24 weeks
Population: Data were collected as a part of main phase of the study only.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pilot: Insulclock Without Feedback (Group A): Participants use the Insulclock and receive daily information on their smartphone on insulin administration (time and dosing) as well as reminders in the event of missing doses. During the study period, information is collected on problems with connectivity, malfunction or any problem with the Insulclock® device.
Arm/Group | Insulclock With Feedback (Group A) | Insulclock Without Feedback (Group B) | Pilot: Insulclock Without Feedback (Group A) | Pilot: Insulclock Without Feedback (Group B)
Number analyzed (Participants) | 40 | 40 | 0 | 0
score on a scale | 15.45 (3.7) | 15.18 (3.05) |  |

4. Secondary Outcome: Change in Diabetes Related Quality of Life (DRQoL) Scores.
Description: DRQoL is a composite score, consisting of a standardized and unweighted Insulin Treatment Experience Questionnaire Score (ITEQ), and Problem Areas in Diabetes (PAID) questionnaire score. ITEQ includes 7 domains: leisure activities (4 items), psychological barriers (2 items), handling (5 items), diabetes control (6 items), dependence (5 items), weight control (3 items), sleep (2 items); + 1 additional item assigned to assess overall satisfaction with current insulin therapy regimen. The PAID contains 20 items that describe negative emotions related to diabetes commonly experienced by patients with diabetes. Each question has five possible answers with a value from 0 to 4, with 0 representing "no problem" and 4 "a serious problem". The scores are added up and multiplied by 1.25, generating a total score between 0 - 100.
Time Frame: Baseline, 24 weeks
Population: The questionnaire was considered originally for use in the study, but no replies were received in a timely manner from the companies in charge of providing licensing for it. Therefore, data was not collected.
Arm/Group | Insulclock With Feedback (Group A) | Insulclock Without Feedback (Group B) | Pilot: Insulclock Without Feedback (Group A) | Pilot: Insulclock Without Feedback (Group B)
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Change in Mean HbA1c.
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the three-month average plasma glucose concentration. The test is limited to a three-month average because the lifespan of a red blood cell is four months (120 days). Change in mean HbA1cas will be measure and recorded to monitor glycemic control.
Time Frame: Baseline, 24 weeks
Population: Data were collected as a part of main phase of the study only.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulclock With Feedback (Group A) | Insulclock Without Feedback (Group B) | Pilot: Insulclock Without Feedback (Group A) | Pilot: Insulclock Without Feedback (Group B)
Number analyzed (Participants) | 40 | 40 | 0 | 0
mg/dL | -0.9 (2.02) | -0.73 (2) |  |

6. Secondary Outcome: Number of Episodes of Hypoglycemia.
Description: Number of episodes of hypoglycemia will be recorded. For this study, symptomatic hypoglycemia is defined as an event with typical symptoms (i.e., sweating, palpitation, and feeling of hunger) with or without confirmation by plasma glucose <54 mg/dl (3.9 mmol/L).
Time Frame: Week 0 through week 24.
Population: Data were collected as a part of main phase of the study only.
Measure: Number; unit: number of events
Arm/Group | Insulclock With Feedback (Group A) | Insulclock Without Feedback (Group B) | Pilot: Insulclock Without Feedback (Group A) | Pilot: Insulclock Without Feedback (Group B)
Number analyzed (Participants) | 40 | 40 | 0 | 0
number of events | 29 | 25 |  |

7. Secondary Outcome: Number of Episodes of Severe Hypoglycemia.
Description: Number of episodes of severe hypoglycemia will be recorded.Severe hypoglycemia is defined as episodes necessitating assistance and associated with measured plasma glucose < 40 mg/dl (2.2 mmol/L), or with prompt recovery after administration of carbohydrates, glucagon, or other resuscitative actions.
Time Frame: Week 0 through week 24.
Population: Data were collected as a part of main phase of the study only.
Measure: Number; unit: number of events
Arm/Group | Insulclock With Feedback (Group A) | Insulclock Without Feedback (Group B) | Pilot: Insulclock Without Feedback (Group A) | Pilot: Insulclock Without Feedback (Group B)
Number analyzed (Participants) | 40 | 40 | 0 | 0
number of events | 1 | 1 |  |

8. Secondary Outcome: Change in Daily Fasting Glucose Profile Averages.
Description: Daily fasting glucose profile averages will be recorded to monitor glycemic control.
Time Frame: Week 0 through week 24.
Population: Data were collected as a part of main phase of the study only.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulclock With Feedback (Group A) | Insulclock Without Feedback (Group B) | Pilot: Insulclock Without Feedback (Group A) | Pilot: Insulclock Without Feedback (Group B)
Number analyzed (Participants) | 40 | 40 | 0 | 0
mg/dL | 142.24 (32) | 146.54 (39) |  |

9. Secondary Outcome: Change in 7-point Self Monitoring of Blood Glucose (SMBG) Profile.
Description: SMBG refers to home blood glucose testing for people with diabetes. 7-point SMBG profile include fasting, before meals, 2 hours after meals, and bedtime.
Time Frame: 3 to 5 days prior to randomization, up to 24 weeks.
Population: Data was only collected at baseline, but not at other visits, therefore it was not possible to assess any change, and it was excluded from the analysis.
Arm/Group | Insulclock With Feedback (Group A) | Insulclock Without Feedback (Group B) | Pilot: Insulclock Without Feedback (Group A) | Pilot: Insulclock Without Feedback (Group B)
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Change in Diabetes Quality of Life Clinical Trial Questionnaire-Revised (DQLCTQ-R) Score
Description: The DQLCTQ-R is a 57-item scale that comprises 8 dimensions: physical function, energy/fatigue, health distress, mental health, satisfaction, treatment satisfaction, treatment flexibility, and frequency of symptoms.
Time Frame: Baseline, 24 weeks.
Population: The questionnaire was considered originally, but no replies were received in a timely manner from the company in charge of providing licensing for it. Therefore, data were not collected.
Arm/Group | Insulclock With Feedback (Group A) | Insulclock Without Feedback (Group B) | Pilot: Insulclock Without Feedback (Group A) | Pilot: Insulclock Without Feedback (Group B)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Insulclock With Feedback (Group A) | Insulclock Without Feedback (Group B) | Pilot: Insulclock With Feedback (Group A) | Pilot: Insulclock Without Feedback (Group B)
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/11 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/40 | 4/40 | 0/11 | 0/7
Other Adverse Events (participants affected / at risk) | 8/40 | 13/40 | 0/11 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulclock With Feedback (Group A) (N=40) | Insulclock Without Feedback (Group B) (N=40) | Pilot: Insulclock With Feedback (Group A) (N=11) | Pilot: Insulclock Without Feedback (Group B) (N=7)
Stroke (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart Failure Readmission (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Surgical Procedures (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulclock With Feedback (Group A) (N=40) | Insulclock Without Feedback (Group B) (N=40) | Pilot: Insulclock With Feedback (Group A) (N=11) | Pilot: Insulclock Without Feedback (Group B) (N=7)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Epigastric pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglicemia (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Toe injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chest pain of muscular etiology (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leg swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non serious work related muscular injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
CHF shortness of breath (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT03224234/Prot_SAP_000.pdf